CLINICAL TRIAL: NCT06664138
Title: Comparison of Remimazolam and Etomidate As Induction Agents for Electroconvulsive Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeongseok Yun (Other)
Responsible Party: Sponsor-Investigator, Yeongseok Yun, Principal Investigator at Dankook University, Dankook University
Organization: Dankook University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DKUH 2023-02-005-002
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Schizophenia Disorder; Major Depression Disorders; Schizoaffective Disorder; Bipolar
MeSH Terms: conditions — Psychotic Disorders | interventions — remimazolam; Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Etomidate & Remimazolam (Other): Patients will receive both etomidate and remimazolam once each to compare their effects while minimizing individual differences in response to the medications. Group E will use etomidate first, followed by remimazolam in the subsequent session.
  Interventions: Drug: Remimazolam; Drug: Etomidate
- Group Remimazolam & Etomidate (Other): Patients will receive both etomidate and remimazolam once each to compare their effects while minimizing individual differences in response to the medications. Group R will use remimazolam first, followed by etomidate in the subsequent session.
  Interventions: Drug: Remimazolam; Drug: Etomidate

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is a recently approved medication used for the induction of general anesthesia and maintenance of sedation. There have been no prior studies using remimazolam for the induction of anesthesia in ECT, and this research aims to investigate the feasibility of using remimazolam as an induction agent for ECT.
Drug: Etomidate — Etomidate is widely used in ECT due to its rapid onset, stable hemodynamic profile, and quick recovery. In this study, remimazolam will be used as the experimental group, while etomidate will serve as the control group.

SUMMARY:
The goal of this clinical trial is to find if patients would awaken quickly after electroconvulsive treatment when remimazolam is used compared to etomidate. It will also learn about the efficacy of remimazolam. The main questions it aims to answer are:

Will using remimazolam as an induction agent for ECT provide sufficient therapeutic effects? Additionally, when compared to etomidate, will remimazolam lead to a quicker return of spontaneous respiration and faster eye opening after the seizure?

Participants will:

Remimazolam and etomidate will be used in a random order, each administered once for the induction of anesthesia in ECT.

Blood pressure, heart rate, and other vital signs will be monitored during the treatment, and the duration of the seizure as well as the shock energy used to induce the seizure will be recorded.

DETAILED DESCRIPTION:
Patients who underwent ECT under general anesthesia between April 2023 and January 2024 were included. The exclusion criteria were as follows: (1) American Society of Anesthesiologists Physical Status ≥3; (2) age <18 or >70 years; and (3) patients with cognitive impairments, such as dementia or delirium. The study sample comprised 30 patients aged 18-70 years who were scheduled to undergo ECT for major depression, schizophrenia, and schizoaffective disorder. The sample size was calculated using G*Power to compare the recovery times between the two groups. On the basis of an effect size of 0.7 obtained from a previous pilot study and a significance level of 0.05, investigators derived a total sample size of 28. Considering a follow-up loss rate of approximately 10%, investigators designed the study to include a total of 30 participants.

The patients were divided into two groups of 15 each and randomly assigned to ei-ther group E or group R using a computer-generated random number table. To minimize variability in recovery speed and response to medication between individuals, investigators devised a crossover study design in which etomidate and remimazolam were administered alternately, with each drug administered once. Patients in group E received etomidate as the induction agent for the first ECT session, followed by remimazolam for the second ECT session a few days later. Conversely, patients in group R received remimazolam as the induction agent for the first ECT session and etomidate for the second ECT session a few days later. The patients and raters were blinded to the administered anesthetic drugs. Blinding was implemented using opaque sealed envelopes that were sequentially numbered.

ECT was conducted following the international standards approved by our institu-tion, using the SpECTrum 5000 Q device (MECTA Corporation, Lake Oswego, OR, USA).

No premedication was administered, and all patients were required to maintain nil per os for at least 8 h before the procedure. During each ECT session, all patients un-derwent non-invasive blood pressure measurement, electrocardiogram, and peripheral oxygen saturation (SpO2) monitoring, and received preoxygenation through an O2 facial mask before anesthesia.

For neuromuscular blockade, succinylcholine (0.8-1.2 mg/kg IV) was used. The an-esthetic dosages were etomidate at 0.15-0.20 mg/kg IV and remimazolam at 0.12-0.15 mg/kg IV. Following admission and monitoring of the patient, preoxygenation was per-formed until SpO2 reached 100%. Then, the induction agent, either etomidate or remi-mazolam, was administered, immediately followed by 100 mcg of remifentanil. Once the patient stopped responding on being called, a cuff was placed on one arm and inflated until the radial artery pulse was no longer detectable. After isolating one arm, succinyl-choline was administered and sufficient time was allowed for fasciculation to resolve before proceeding. After adequate time for the muscle relaxant to take effect, electrical currents were delivered to the brain through electrodes placed on the scalp. The intensity of the current was determined according to an established psychiatric protocol, and in the absence of a seizure, was increased by 10 J in three successive attempts. If a seizure lasting longer than 30 s was induced, the treatment was considered successful. The duration of the seizure and corresponding shock intensity were recorded for each patient.

Following the seizure, mask ventilation was continued until spontaneous respiration returned. The time from the end of the seizure until the patient's spontaneous tidal volume reached ≥200 mL was measured and defined as the self-respiration recovery time. Additionally, the time from the end of the seizure until the patient opened their eyes spontaneously, either in response to a gentle tap or verbal stimulation, was measured and defined as the eye-opening recovery time.

Apart from the induction agent, there were no differences between the two groups in terms of procedural techniques, anesthetic management during surgery, or cardiovascular support.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years
* Patients diagnosed with major depression, schizophrenia, and schizoaffective disorder who are scheduled to undergo ECT treatment

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status ≥3
* Age <18 or >70 years
* Patients with cognitive impairments, such as dementia or delirium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Self respiration recovery time | From enrollment to the end of treatment at one week
  After the induction of anesthesia, a shock is administered to induce a seizure. The time is measured from the end of the seizure until the patient's spontaneous tidal volume exceeds 200 ml.
eye opening recovery time | From enrollment to the end of treatment at one week
  After the induction of anesthesia, a shock is administered to induce a seizure. The time is measured from the end of the seizure until the patient's spontaneous eye opening.

SECONDARY OUTCOMES:
Mean Blood pressure | From enrollment to the end of treatment at one week
  Mean Blood pressure measured using non-invasive blood pressure, immediately after induction, immediately after shock, and at awakening state, with measurements taken in mmHg
Heartrate | From enrollment to the end of treatment at one week
  Heartrate measured using electrocardigram, immediately after induction, immediately after shock, and at awakening state, with measurements taken in bpm(beats per minute)
seizure duration | From enrollment to the end of treatment at one week
  The duration of the induced seizure following the administration of the shock, with measurements taken in seconds
shock energy | From enrollment to the end of treatment at one week
  The amount of energy delivered by the shock used to induce the seizure with the ECT machine, measured in Joules.

CONTACTS AND LOCATIONS:
Locations (1):
- Dankook University Hospital, Cheonan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
All data generated during the study will be shared and can only be provided to individuals with academic purposes, excluding any personal information about the patients, upon request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code